CLINICAL TRIAL: NCT06405503
Title: Impact of Primary Language on Treatment and Outcomes in Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: Bristol-Myers Squibb (Industry); Yale University (Other)
Responsible Party: Principal Investigator, Linda Anne Feagins, MD, Associate Professor of Medicine, University of Texas at Austin
Other Study IDs: STUDY00004331
Record Dates: First submitted 2023-04-10; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- English as primary language
  Interventions: Other: NO INTERVENTION
- Non-English as primary language
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION - OBSERVATIONAL ONLY

SUMMARY:
A thorough discussion of treatment options to manage inflammatory bowel disease (IBD), including the risks and benefits of each class of medication, can be a complex discussion and time consuming. Having to use a translator adds an additional layer of time and complexity to these discussions as well as potential misunderstanding. Further, in addition to language, cultural differences can also play into treatment acceptance.

This study aims to determine the impact of primary language on the selection of treatment for IBD and on disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Confirmed diagnosis of IBD (CD, UC or indeterminate colitis)
* Willing to provide consent for participation
* Managed at an outpatient clinic either the Yale New Haven Hospital system or the University of Texas at Austin Hospital system.

Exclusion Criteria:

* Patients <18
* No confirmed diagnosis of IBD
* Not planning to continue care at either study site (i.e. presenting for a consultation only)
* Unwilling to provide signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target population will include adult subjects (ages 18 and older) with confirmed IBD who do and do not identify English as their primary language. These subjects will be either new or returning patients seen in the outpatient clinics at either the Yale New Haven Hospital system or the University of Texas at Austin affiliated hospitals or clinics. Men and women and persons of all races and ethnicities will be encouraged to participate in an equal basis.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Current use of advanced therapy | baseline
  Use of or prescription of a biologic or small molecule therapy to treat inflammatory bowel disease

SECONDARY OUTCOMES:
IBD-related disease complications | 6 months
IBD-related disease complications | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School at the University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided